CLINICAL TRIAL: NCT06548152
Title: AQUALIS: Quality of Life of Patients With Chronic Lymphocytic Leukemia Treated With Acalabrutinib in France: a Retrospective Observational Study Based on Data Extracted From the PLATON Database
Brief Title: AQUALIS:QoL of CLL Patients Treated With Acalabrutinib in France, Retrospective Study Based on Data From PLATON Database
Acronym: AQUALIS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Hospitalidee (Unknown); Hospitalidee has been asserted to be a valid organization name by UHToulouse (Unknown)
Responsible Party: Sponsor
Other Study IDs: D8220R00057
Record Dates: First submitted 2024-07-17; First posted 2024-08-12 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia (LLC); Quality of life; Acalabrutinib; France; Retrospective observational study; PLATON database
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
QoL is often not assessed in real-world studies; hence, there is limited understanding about the real-world QoL of patients diagnosed with CLL. Besides, studies evaluating QoL have largely focused on comparing treated and untreated populations. In particular, QoL of patients treated with acalabrutinib has not been evaluated in a real-life setting.

The aim of this study is to describe the QoL of CLL patients treated with acalabrutinib between the treatment initiation and twelve months after, in a real-life setting.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS

Background/Rationale:

CLL is the most prevalent leukemia among adults. The estimated incidence of CLL was 4 674 in 2018 in France, 59% in men with a median age of 71 in men and 73 in women. 95% of patients are older than 51 yrs at diagnosis. 5-yr survival is above 89% for patients diagnosed between 2010 and 2015. Yet, CLL cannot be cured. Some patients will require monitoring while others need to be treated. Treatment is based on both chemo-immunotherapies (CIT) and target therapies. Treatment choice depends on several parameters: age, patient general condition, comorbidities, prognostic factors, cytogenetic status. CIT have shown to improve overall survival (OS). Targeted therapies have changed the management and offer treatment options among older patients and those with comorbidities who have unacceptable side effects with CIT. Acalabrutinib (also known as ACP-196 and Calquence®), is a selective and irreversible small molecule inhibitor of BTK. Authorized as 1st or 2nd line treatment in France in November 2020. Its safety and efficacy were explored in phase III clinical trials ELEVATE-TN, ASCEND, and ELEVATE-R/R. Because CLL is, by definition, a chronic disease and requires long-term treatment and because many patients have comorbidities, it is essential to consider quality of life (QoL) of patients.14 In addition, the condition itself substantially impacts QoL.Patients with CLL experienced worse QoL than the general population across several domains, including symptoms (e.g. fatigue and sleep disturbances), as well as physical and mental functioning. Acalabrutinib has shown great efficacy associated with a good safety profile in clinical trials11,12,14. Moreover, it is an oral treatment that does not require intravenous injections when taken as monotherapy. This treatment modality associated with the favorable safety profile of acalabrutinib could have a positive impact on the QoL of patients. Indeed, patients could continue to live a normal life at home, surrounded by their relatives. QoL is often not assessed in real-world (RW) studies; hence, there is limited understanding about the RW QoL of patients diagnosed with CLL. Besides, studies evaluating QoL have largely focused on comparing treated and untreated populations. In particular, QoL of patients treated with acalabrutinib has not been evaluated in a real-life setting. The aim of this study is to describe the QoL of CLL patients treated with acalabrutinib between the treatment initiation and 12 months after, in a real-life setting.

Objectives:

Primary Objective : To measure QoL score of CLL patients treated with acalabrutinib, from treatment initiation and up to 12 months -Overall scores and scores in each domain of QoL questionnaires (EORTC-QLQ-C30 ) at acalabrutinib treatment initiation and at 3, 6, 9 and 12 months after initiation -Proportion of patients with an increase, a decrease, or no change in QoL scores over time (between each time point) Main Secondary Objectives: To describe QoL and precisely the level and evolution of all symptoms -Patients demographics (age, gender…) at acalabrutinib treatment initiation -Clinical characteristics at acalabrutinib treatment initiation (CLL diagnosis, Binet classification, comorbidities of interest) -Clinical characteristics quarterly up to 12 months (disease status) -Score is calculated with standardized EORTC-CLL17 questionnaire At acalabrutinib treatment initiation and at 3, 6, 9 and 12 months after initiation To measure the evolution of observance -Score is calculated with standardized GIRERD grid at 3, 6, 9 and 12 months after initiation To describe treatment patterns in CLL patients treated with acalabrutinib, overall and by age group -Acalabrutinib treatment: line, monotherapy or with obinutuzumab, posology, duration, reason for discontinuation if any To describe participating sites characteristics -Type of physician practice (public/private/mixed) -Type of care structure (CHU/ CHG…) -Existing patient support program (yes/no, type) Methods: Study design: This is a retrospective, observational study focusing on the QoL and experience of CLL patients treated with acalabrutinib in France in a real-life setting. This study is using secondary data of patients included in the national multicenter longitudinal cohort PLATON (sponsor HOSPITALIDEE) (clinical trial registration N° 2023-A01569-36). This cohort is enrolling patients with hematological malignancies including CLL patients. A follow-up of 12 months from initial cancer diagnosis / or patient enrollment is planned in the PLATON study. The current AQUALIS study mainly aims at describing CLL patient QoL and experience from acalabrutinib initiation, quarterly and up to 12 months post initiation. Patient and disease characteristics, treatment patterns, disease status over time will also be described. Thus, the patient population eligible for entering the AQUALIS study will be treatment naïve CLL patients enrolled in the PLATON study and having initiated acalabrutinib, at the time of data extraction. Only patients with a full T0 will be considered as included. Several data extraction from PLATON database and data cut-off are planned to address AQUALIS study objectives and planned publication plan. No extra-visit, nor specific additional examination nor intervention are required for patients eligible to enter the AQUALIS study. Data to be extracted and analyzed will be exclusively those already recorded in the PLATON database. HOSPITALIDEE will insure that in each center participating to PLATON cohort, all patients fulfilling the PLATON eligibility criteria have been informed about the PLATON study before being enrolled in the PLATON database and do not object to secondary use of their data. The AQUALIS study does not involve human person according to the French legislation. Data Source(s): The AQUALIS study will be a secondary use of data issued from the French PLATON cohort. The PLATON cohort is a national prospective cohort enrolling patients diagnosed with malignant hemopathies, aiming at to offer personalized information to patients to improve their QoL and guide their use of complementary care. PLATON is designed to ensure patients follow-up in the long term and on a European scale. This project is sponsored by HOSPITALIDEE and coordinated by Loic Raynal under the scientific responsibility of Pr Loïc Ysebaert. The sponsor has been granted with appropriate regulatory and ethics local approvals for the conduct of the study. Patients eligible to PLATON are informed about the study and are requested to sign a specific informed consent if they do agree for participation and for their data being processed. It is planned that 120 patients are enrolled and followed-up to 12 months from enrollment. Data are collected at patient inclusion, and on a regular basis (every 3 months) during the follow-up, according to routine practice. Socio-demographic, clinical, biological data, treatments patterns, etc..(Pathology, treatments, history, lifestyle, sociodemographic analysis, patient profile, preferences…) are collected via an electronic data capture tool and hosted in a centralized securized data center. Patient QoL and experience is also collected at 5 timepoints using 4 questionnaires . The PLATON database is managed by HOSPITALIDEE using their own software. A data-management plan and a consistency check program were established during database development. Quality controls of the data are performed: i) automatic data consistency check; ii) data management control through regular sending of queries; iii) regular e-control of entered data by the project manager; iv) remote and / or on-site data monitoring of at least 100% of the data entered. Data collection and hosting, data management, and statistical analysis of PLATON data are handled by HOSPITALIDEE. No patient-level data will be transmitted to AstraZeneca. Only aggregated data will be delivered, based on the current AQUALIS protocol and a related statistical analysis plan. Study population The AQUALIS study population will be a subgroup of patients enrolled in PLATON database following inclusion and exclusion criteria as described below.

Inclusion-Exclusion criteria: please see details in "ELIGIBILITY" SECTION. Outcome(s): Please see details "OUTCOME MEASURES" SECTION.

Patient study questionnaires :

In our research protocol, we have chosen the EORTC QLQ-C30 as our primary tool for evaluating quality of life. To address the potential overlap with the MD Anderson Symptom Inventory (MDASI), we have substituted the MDASI with the QLQ-CLL17, a supplementary module to the QLQ-C30 specifically designed for chronic lymphocytic leukemia. This addition enhances the relevance and specificity of our study's context. Alongside the QLQ-C30, the QLQ-CLL17 provides a comprehensive assessment tailored to our research objectives. Furthermore, we have opted to use neither FACIT-TS-G questionnaire nor the Cancer Therapy Satisfaction Questionnaire (CTSQ). Our decision was influenced by concerns about redundancy and the length of these questionnaires, which could potentially burden respondents and affect the quality of the data collected. This decision was also rooted in the observation that the measurement of satisfaction is conducted in a notably heterogeneous manner across existing questionnaires, lacking a standard, and only partially covering the scope of satisfaction. This perspective was shared by several hematologists we collaborate with, including Loïc Ysebaert, who notes that to date, no satisfaction questionnaire has become the reference.

While it's possible to publish using any questionnaire, the main goal of our protocol and studies conducted through Platon is to utilize standardized instruments like the QLQ-C30, allowing for the comparison of results. However, satisfaction with treatment serves as an illuminating indicator, rather than a comparative outcome to judge the superiority of patients' quality of life. It is more of an "insight". This view is endorsed by the Aqualis scientific committee, with whom we co-developed the satisfaction questionnaire. Based on patient feedback and scientific committee recommendations, we have created a simplified, non-standardized version to more effectively capture treatment satisfaction, prioritizing the relevance and comfort of our participants in the data collection process.

The aim is to ensure the highest possible completion rate over time, from T0 to T12. The questionnaire we have implemented is inspired by the CTSQ, featuring questions on the patient's overall satisfaction, the impact of their treatment on daily life, the occurrence of adverse effects and their impact (with a disclaimer directing to the adverse effect reporting portal), and the potential use of support care services.

Additionally, the Girerd questionnaire will help monitoring treatment adherence, providing valuable insights into how patients comply with their prescribed regimens.

Sample Size Estimations: - Given the observational nature of the study and the descriptive nature of the primary objective, no pre-defined hypothesis testing is expected to be used to address the primary objective. - Assuming a 20% loss of follow-up, the number of patients to address the exploratory objective will be 120*0.8=96. Statistical Analysis: With a sample size of 120 patients (treated with acalabrutinib as a first-line therapy), we will have enough power to detect a change (including an improvement) in the QoL of patients over time with one QoL (EORTC-QLQ-C30). A comprehensive statistical analysis plan (SAP) will be developed before the first analysis and finalized before the database lock. A descriptive analysis will be conducted on all variables for which data have been extracted for the overall study population and sub-groups of interest. Continuous, quantitative, variable summaries will include: the number of patients (N) (with non-missing values), mean, standard deviation (SD), median, minimum, maximum, 1st, and 3rd quartiles. Categorical, qualitative, variables summaries will include the frequency and percentage of patients per category. The denominator for percentage calculations will be based on the number of observed data, unless otherwise specified. All applicable statistical tests will be two-sided and will be performed at a 5% significance level. Missing values will not be imputed. Results will be presented overall and by treatment line and by age group, as specified in the study objectives. Additional subgroups of interest may be further investigated and discussed in the protocol and/or the SAP.

ELIGIBILITY:
Inclusion criteria:

The following patients will be eligible for inclusion in the AQUALIS study :

* Patient enrolled in the PLATON database
* Patient ≥18 years old
* Treatment naïve CLL patient treated with acalabrutinib in a real life setting. Treatment pattern is Acala mono or Acala + Obinutuzumab
* Patient who do not object to his health data collected in PLATON study being re-use for analysis/research purpose
* Patients who started Acala but discontinued before 12 months are also included.

Exclusion criteria:

* Pregnant women
* Patients under protection of justice
* Patients over the age of 18 and unable to express their non-opposition
* Patients with prior CLL treatments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be a subgroup of patients enrolled in PLATON database as described below.
  Inclusion criteria:
  The following patients will be eligible for inclusion :
  * Patient enrolled in the PLATON database
  * Patient ≥18 years old
  * Treatment naïve CLL patient treated with acalabrutinib in a real life setting. Treatment pattern is Acala mono or Acala + Obinutuzumab
  * Patient who do not object to his health data collected in PLATON study being re-use for analysis/research purpose
  * Patients who started Acala but discontinued before 12 months are also included.
  Exclusion criteria:
  * Pregnant women
  * Patients under protection of justice
  * Patients over the age of 18 and unable to express their non-opposition
  * Patients with prior CLL treatments
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To measure QoL score of CLL patients treated with acalabrutinib, from treatment initiation and up to 12 months | From treatment initiation and up to 12 months
  * Overall scores and scores in each domain of QoL questionnaires (EORTC-QLQ-C30 ) at acalabrutinib treatment initiation and at 3, 6, 9 and 12 months after initiation
  * Proportion of patients with an increase, a decrease, or no change in QoL scores over time (between each time point)

SECONDARY OUTCOMES:
To describe QoL and precisely the level of all symptoms | Treatment initiation
  * Patients demographics at acalabrutinib treatment initiation
  * Clinical characteristics at acalabrutinib treatment initiation
To describe QoL and precisely the level and evolution of all symptoms | From treatment initiation and up to 12 months
  * Clinical characteristics quarterly up to 12 months
  * Score is calculated with standardized EORTC-CLL17 questionnaire At acalabrutinib treatment initiation and at 3, 6, 9 and 12 months after initiation
Data outcomes analyze and link together | From treatment initiation and up to 12 months
  The severity of symptoms and the interference with daily living caused by these symptoms will be assessed using EORTC QLQ-CLL17 questionnaire. The overall scores of the QLQ-CLL17 questionnaire will be presented: at acalabrutinib treatment initiation and at 3, 6, 9 and 12 months after initiation.
  A mixed model will be used on repeated measurements of total QLQ-CLL17 score to study the evolution of QLQ-CLL17 after acalabrutinib treatment initiation. The model will be adjusted on age and sex and time of measurement as fixed effect.
  Disease status will be described quarterly up to 12 months after treatment initiation according to the following status:
  -missing value (patients not followed or missing score), complete response, partial response, partial response with lymphocytosis, stable disease, progressive disease Disease status will be analysed according to a sunburst diagram and a Sankey diagram.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Saint-Affrique, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/